CLINICAL TRIAL: NCT02124681
Title: Rediscovering Hydroxychloroquine as a Novel Insulin Sensitizer
Acronym: REHNIS
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Responsible Party: Principal Investigator, Frederico Toledo, Associate Professor, University of Pittsburgh
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: PRO13060248
Record Dates: First submitted 2014-04-24; First posted 2014-04-28 (Estimated); Last update posted 2017-06-06 (Actual); Status verified 2017-06

CONDITIONS: Insulin Resistance
MeSH Terms: conditions — Insulin Resistance | interventions — Hydroxychloroquine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Placebo (Placebo Comparator): Placebo PO
  Interventions: Other: Placebo
- Hydroxychloroquine (Experimental): Hydroxychloroquine sulfate 400mg PO QD
  Interventions: Drug: Hydroxychloroquine

INTERVENTIONS:
Drug: Hydroxychloroquine — Hydroxychloroquine sulfate 400mg/d PO for 13±1 weeks
  Arms: Hydroxychloroquine
Other: Placebo — Placebo PO for 13±1 weeks
  Arms: Placebo

SUMMARY:
Current options to treat insulin resistance in diabetes are fairly limited. For this reason, novel treatments would represent a major progress. The generic drug hydroxychloroquine (HCQ) has poorly understood effects on blood sugar metabolism. In this study, the investigators will examine the mechanisms by which this drug affects glucose metabolism and which cells are affected. Findings emanating from this project will help establish whether HCQ may be a viable treatment for disorders of glucose metabolism.

ELIGIBILITY:
Inclusion Criteria:

* Age 21-69 years-old;
* BMI 28-40;
* Presence of at least one of the following markers of insulin resistance: a) fasting hyperinsulinemia (>7 uU/ml by ultrasensitive insulin assay); impaired fasting glucose (100-125 mg/dl); prior history of impaired glucose tolerance provided by the participant; history of previous gestational diabetes; history of PCOS; waist circumference >40" (men) or >35" (women) (cut-offs from ATP-III criteria for metabolic syndrome).

Exclusion Criteria:

* Pregnancy, or unable/unwilling to avoid pregnancy during the study;
* Unstable cardiopulmonary disease, hepatitis, liver dysfunction, renal insufficiency, or any other medical condition affecting glucose metabolism or safety during the study;
* Diabetes;
* Medications that affect glucose metabolism: (e.g. systemic glucocorticoids, antipsychotics);
* History of hypersensitivity to local lidocaine, similar anesthetics, or HCQ;
* History of G6PDH deficiency;
* History of retinopathy;
* Weight instability (>3Kg of weight change in the past three months);
* Bariatric surgery in the last two years, intention to lose weight or engage in exercise regimen during study;
* Alcohol intake >1 drink/day (averaged);
* Hemoglobin <10g%

Ages: 21 Years to 69 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2014-04; Primary Completion 2016-08 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
Insulin sensitivity in muscle and liver | 13±1 weeks

SECONDARY OUTCOMES:
biomarkers of inflammation | 13±1 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Frederico Toledo, MD, Principal Investigator — University of Pittsburgh
Locations (1):
- UPMC Montefiore Hospital, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No